CLINICAL TRIAL: NCT00002295
Title: A Double-Blind Placebo-Controlled Study to Investigate the Action of Isoprinosine (Inosiplex) in Patients With Severe Acquired Immunodeficiency Syndrome
Brief Title: A Study of Isoprinosine in Patients With Severe AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newport Pharmaceuticals International (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 008F; ISO-141-USA
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-06

CONDITIONS: HIV Infections
Keywords: Infusions, Intravenous; Drug Evaluation; Administration, Oral; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Biological Availability
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Inosine Pranobex

INTERVENTIONS:
Drug: Inosine pranobex

SUMMARY:
To evaluate the effect of Isoprinosine in patients diagnosed as having AIDS relative to:

Laboratory (immunologic defects):

* Comparison of total helper and suppressor T-cell numbers among the groups.
* Comparison of changes in natural killer cell activity.
* Comparison of other laboratory findings among the groups.

Clinical changes:

* Comparison of the frequency of opportunistic infections among the groups.
* Comparison of the frequency of the development of AIDS-related malignancies.
* Comparison of other clinical manifestations relative to severity and time of onset.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with a history of gout, urolithiasis, nephrolithiasis, renal dysfunction, and severe gastric ulcer are excluded.

Concurrent Medication:

Excluded:

* Steroids.
* Cytotoxic immunosuppressive agents.
* Radiotherapy.

The following are excluded:

* Critically ill patients.
* Patients receiving steroids, cytotoxic immunosuppressive agents, radiotherapy.
* Patients who have received any other immunotherapy.
* Patients with a history of gout, urolithiasis, nephrolithiasis, renal dysfunction, and severe gastric ulcer.

Prior Medication:

Excluded:

* Any other immunotherapy.

Patients with severe AIDS and specified laboratory immunologic defects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Newport Pharmaceuticals International Inc, Laguna Hills, California, United States